CLINICAL TRIAL: NCT03919448
Title: A Double-blind, Randomized, Balanced, Parallel Group, Phase I Study Comparing Pharmacokinetics and Safety of Bevacizumab
Brief Title: A Phase I Study Comparing Pharmacokinetics and Safety of Bevacizumab
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Laboratorios Richmond S.A.C.I.F. (Industry)
Collaborators: FP Clinical Pharma S.R.L. (Industry); Syngene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 0221
Record Dates: First submitted 2019-04-15; First posted 2019-04-18 (Actual); Results first posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2022-08

CONDITIONS: Pharmacokinetics; Safety Issues
Keywords: Bevacizumab; Biosimilar; Antineoplastic Agents; Bioequivalence; Immunogenicity; safety; healthy male volunteers
MeSH Terms: interventions — Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Zutrab® (Bevacizumab Richmond) (Active Comparator): a single 1 mg/kg IV dose of Bevacizumab
  Interventions: Biological: Bevacizumab
- Avastin® (Active Comparator): a single 1 mg/kg IV dose of Bevacizumab
  Interventions: Biological: Bevacizumab
- Cizumab® (Active Comparator): a single 1 mg/kg IV dose of Bevacizumab
  Interventions: Biological: Bevacizumab

INTERVENTIONS:
Biological: Bevacizumab — Single-dose infusion

SUMMARY:
The aim of the Clinical study is to evaluate the pharmacokinetic and safety profile of a new formulation of Bevacizumab (Zutrab®, Argentinian origin) when compared to two already marketed formulations of Bevacizumab Avastin® (reference product) and Cizumab® (Indian origin), to establish similarity.

DETAILED DESCRIPTION:
Three-way bridge phase 1 trial. It is conducted in healthy, male adult subjects, it is single-dose, double-blind, parallel groups, randomized and balanced.

Blood samples are collected for up to 90 days, to determine serum drug concentration and anti-drug antibodies. Safety and tolerability are also assessed.

ELIGIBILITY:
Inclusion Criteria:

* Study subjects must be willing and able to provide written informed consent
* Subjects of study, volunteers, adults, healthy.
* Study subjects whose safety and complementary laboratory tests are within normal values or which, in the Investigator's opinion, do not have clinical relevance: blood count, erythrosedimentation, hepatogram, urea, creatinine, glucose, coagulogram, serology for HIV, hepatitis B , hepatitis C, complete urinalysis, detection of drugs of abuse in urine and electrocardiogram.
* Sample taken for immunogenicity
* Body mass index between 19 and 27 kg / m2 at the screening visit.
* Subjects of study preferably non-smokers.
* Men with a partner of childbearing age must agree that their partner uses an adequate contraceptive method before entering the study and for at least 3 months after the end of the study. It is understood as a contraceptive method suitable to any hormonal contraceptive method or intrauterine device (which should be established before the start of the study) and the use of a spermicide as a barrier method. The use of a barrier method alone or sexual abstinence is not considered adequate.
* Subjects must agree not to donate sperm during the study and for 4 months after treatment.

Exclusion Criteria:

* History of pulmonary, gastrointestinal, hepatic, renal, hematological, endocrine-metabolic, neurological or psychiatric illnesses (depressive disorders, in particular) at the time of taking the anamnesis and the physical examination during the first visit of the Protocol of Clinical research.
* History of gastrointestinal surgeries (except uncomplicated appendectomy, at least 3 months old).
* History of major surgery, surgical biopsy and / or history of significant trauma within 1 month of the screening visit.
* Specifically, pre-existing gastrointestinal conditions such as abdominal fistulas, gastrointestinal perforation within 6 months of the screening visit.
* Specifically, preexisting gastrointestinal conditions such as acute or subacute intestinal occlusion.
* Specifically, history of inflammatory bowel disease.
* History of hemorrhagic diseases and / or coagulopathies and / or thromboembolic events.
* History of heart and vascular diseases: specifically myocardial infarction, unstable angina, cerebrovascular accident, uncontrolled arterial hypertension and cardiac arrhythmias.
* Background or current history of alcohol or drug abuse.
* Blood donation within 3 months prior to selection.
* Administration of any other drug under investigation or participation in a clinical research trial within 3 months prior to the planned participation in this Clinical Research Protocol.
* History of clinically significant diseases or disorders that, in the opinion of the Investigator, may impede the participation of the study subject for safety reasons or that may influence the results of the same as well as the ability of the study subject to participate in the Clinical Research Protocol.
* History of hypersensitivity to bevacizumab and / or any of the excipients.
* Study subjects who present contraindications to therapy
* Study subjects who have received (2 weeks before) or are receiving aspirin or clopidogrel
* The study subjects must have suspended any pharmacological treatments at least 2 weeks before the initiation of this Clinical Research Protocol.
* Non-cooperative study subjects
* Study subjects employed by the Researcher or the Clinical-Pharmacokinetic Research Unit, with direct participation in the Clinical Research Protocol or other clinical protocols under the Direction of the Researcher or the Clinical-Pharmacokinetic Research Unit
* Physical findings and laboratory analyses:
* Cardiac, pulmonary, gastrointestinal, hepatic, renal, hematological, endocrine-metabolic, neurological disease or psychiatric disorder (depressive disorders, in particular)
* Evidence of ulcers, unhealed wounds or bone fractures.
* Clinically significant abnormalities in any laboratory analysis, and electrocardiogram
* Positive serology for HIV, hepatitis B, hepatitis C

Ages: 21 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-09-11 (Actual); Study Completion 2019-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ethel C Feleder, MD, Principal Investigator — FP Clinical Pharma S.R.L.
Locations (1):
- FP Clinical Pharma S.R.L., Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 112 enrolled participants, 90 met inclusion criteria and were randomized to treatment.
Period: Overall Study
Arm/Group | Zutrab® (Bevacizumab Richmond) | Avastin® | Cizumab®
Started | 30 | 30 | 30
Completed | 29 | 30 | 30
Not Completed | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zutrab® (Bevacizumab Richmond) | Avastin® | Cizumab® | Total
Number analyzed (Participants) | 29 | 30 | 30 | 89
Age, Customized [Count of Participants; unit: Participants]
  21 to 55 years | 29 | 30 | 30 | 89
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 29 | 30 | 30 | 89
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Mass Index (BMI) [Mean (Full Range); unit: kg/m^2] | 24.05 [19.56 to 26.94] | 24.06 [19.01 to 26.99] | 24.85 [19.23 to 26.91] | 24.32 [19.01 to 26.99]

OUTCOME MEASURES:

1. Primary Outcome: Peak Serum Concentration of Bevacizumab (Cmax)
Description: Cmax will be obtained directly from the serum concentration-time curve
Time Frame: 0, 0.33, 0.5, 1, 1.5 hours during infusion, 0.33, 0.66, 1, 2, 4, 8, 12, 24, 48, 72, 96, 120, 168, 336, 504, 672, 840, 1008, 1176, 1344, 1512 hours post-infusion
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Zutrab® (Bevacizumab Richmond) | Avastin® | Cizumab®
Number analyzed (Participants) | 29 | 30 | 30
ng/ml | 22144.83 (5550.07) | 21540 (4382) | 22566.67 (8368.14)
Statistical Analysis 1: Comparison: Zutrab® (Bevacizumab Richmond) vs Avastin®; The null hypothesis (H0) of ANOVA is that there is no difference among group means. The alternate hypothesis (H1) is that at least one group differs significantly from the overall mean of the dependent variable; Test type: Equivalence — The comparable bioavailability was achieved if 90 % confidence intervals (CIs) for the test-to-reference ratios of the geometric means of Cmax, Area Under the Serum Concentration-time Curve of Bevacizumab (ABC0-t) fell within the 80.00-125.00 % acceptance criteria; p = 0.9766, ANOVA — Power of ANOVA: 0,93; Hazard Ratio (HR) = 101.55, 90% CI 2-sided [90.19 to 114.34]
Statistical Analysis 2: Comparison: Avastin® vs Cizumab®; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.9766, ANOVA — Power of ANOVA: 0,93; Hazard Ratio (HR) = 100.95, 90% CI 2-sided [89.75 to 113.55]
Statistical Analysis 3: Comparison: Zutrab® (Bevacizumab Richmond) vs Cizumab®; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — As supplementary information, Test Product 1 vs. Test Product 2 shall also be compared. The comparable bioavailability was achieved if 90 % confidence intervals (CIs) for the test1-to-test2 ratios of the geometric means of Cmax, Area Under the Serum Concentration-time Curve of Bevacizumab (ABC0-t) fell within the 80.00-125.00 % acceptance criteria; p = 0.9766, ANOVA; Hazard Ratio (HR) = 100.59, 90% CI 2-sided [88.16 to 114.77]

2. Primary Outcome: Area Under the Serum Concentration-time Curve of Bevacizumab (ABC0-t)
Description: Area under the serum concentration-time curve from time zero to the last experimental point, will be calculated by the trapezoidal rule
Time Frame: Day 1 to Day 63
Measure: Mean (Standard Deviation); unit: h*ng/ml
Arm/Group | Zutrab® (Bevacizumab Richmond) | Avastin® | Cizumab®
Number analyzed (Participants) | 29 | 30 | 30
h*ng/ml | 5153367.55 (1276468.14) | 5641733.72 (1160626.12) | 5500141.94 (1849362.76)
Statistical Analysis 1: Comparison: Zutrab® (Bevacizumab Richmond) vs Avastin®; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — The comparable bioavailability was achieved if 90% confidence intervals (CIs) for the test to reference ratios of the geometric means of Cmax, Area under the serum concentration-time curve of bevacizumab (ABC0-t) fell within the 80.00-125.00% acceptance criteria; p = 0.3617, ANOVA — Power of ANOVA: 0,95; Hazard Ratio (HR) = 90.82, 90% CI 2-sided [81.21 to 101.57]
Statistical Analysis 2: Comparison: Avastin® vs Cizumab®; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.3617, ANOVA — Power of ANOVA: 0.95; Hazard Ratio (HR) = 94.87, 90% CI 2-sided [84.91 to 105.99]
Statistical Analysis 3: Comparison: Zutrab® (Bevacizumab Richmond) vs Cizumab®; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — [test comment as in outcome 1, analysis 3]; p = 0.3617, ANOVA; Hazard Ratio (HR) = 95.73, 90% CI 2-sided [84.82 to 108.05]

3. Primary Outcome: Area Under the Serum Concentration- Time Curve ob Bevacizumab (ABC0-∞)
Description: Area under the serum concentration- time curve from time zero to infinity
Time Frame: Day 1 to Day 63
Measure: Mean (Standard Deviation); unit: h.ng/ml
Arm/Group | Zutrab® (Bevacizumab Richmond) | Avastin® | Cizumab®
Number analyzed (Participants) | 29 | 30 | 30
h.ng/ml | 5374225.878 (1340507.11) | 5919875.18 (1276082.30) | 5777584.241 (1951347.40)
Statistical Analysis 1: Comparison: Zutrab® (Bevacizumab Richmond) vs Avastin®; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — 80.00-125.00% acceptance criteria; p = 0.3529, ANOVA — Power of ANOVA: 0.94; Hazard Ratio (HR) = 90.46, 90% CI 2-sided [80.64 to 101.47]
Statistical Analysis 2: Comparison: Avastin® vs Cizumab®; Test type: Equivalence — 80.00-125.00% acceptance criteria; p = 0.3529, ANOVA — Power of ANOVA: 0.94; Hazard Ratio (HR) = 95.02, 90% CI 2-sided [84.80 to 106.49]
Statistical Analysis 3: Comparison: Zutrab® (Bevacizumab Richmond) vs Cizumab®; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — [test comment as in outcome 1, analysis 3]; p = 0.3529, ANOVA; Hazard Ratio (HR) = 95.19, 90% CI 2-sided [84.17 to 107.67]

4. Secondary Outcome: Time to Reach the Peak Serum Concentration (Tmax)
Description: Time to reach the peak serum concentration, which will be obtained directly from the serum concentration curve- time
Time Frame: Day 1 to Day 63
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Zutrab® (Bevacizumab Richmond) | Avastin® | Cizumab®
Number analyzed (Participants) | 29 | 30 | 30
h | 9.34 (11.65) | 16.69 (22.79) | 5.64 (7.46)

5. Secondary Outcome: Terminal Elimination Rate Constant (λz)
Description: Terminal elimination rate constant will be calculated by linear regression analysis of the semi-logarithmic curve
Time Frame: Day 1 to Day 63
Measure: Mean (Standard Deviation); unit: 1/h
Arm/Group | Zutrab® (Bevacizumab Richmond) | Avastin® | Cizumab®
Number analyzed (Participants) | 29 | 30 | 30
1/h | 0.002 (0.001) | 0.002 (0.001) | 0.002 (0.001)

6. Secondary Outcome: Elimination Half Life (T1/2)
Description: To assess pharmacokinetic parameters
Time Frame: Day 1 to Day 63
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Zutrab® (Bevacizumab Richmond) | Avastin® | Cizumab®
Number analyzed (Participants) | 29 | 30 | 30
h | 352.19 (173.17) | 344.58 (82.04) | 371.86 (315.65)

7. Secondary Outcome: Systemic Clearance (CL)
Description: To assess pharmacokinetic parameters
Time Frame: Day 1 to Day 63
Population: To asses pharmacokinetic parameters
Measure: Mean (Standard Deviation); unit: ml/h/kg
Arm/Group | Zutrab® (Bevacizumab Richmond) | Avastin® | Cizumab®
Number analyzed (Participants) | 29 | 30 | 30
ml/h/kg | 0.20 (0.05) | 0.18 (0.04) | 0.19 (0.06)

8. Secondary Outcome: Distribution Volume
Description: To assess pharmacokinetic parameters
Time Frame: Day 1 to Day 63
Measure: Mean (Standard Deviation); unit: ml/kg
Arm/Group | Zutrab® (Bevacizumab Richmond) | Avastin® | Cizumab®
Number analyzed (Participants) | 29 | 30 | 30
ml/kg | 99.10 (51.39) | 85.35 (17.62) | 97.91 (67.17)

9. Secondary Outcome: Number of Participants With Positive Anti-bevacizumab Serum Antibodies Detection
Description: To assess the immunogenic potential of the products under investigation, samples were taken for the determination of anti-bevacizumab serum antibodies for each randomized volunteer subject.
Time Frame: Screening and end of study (Day 63)
Measure: Number; unit: participants tested positive for ADA
Arm/Group | Zutrab® (Bevacizumab Richmond) | Avastin® | Cizumab®
Number analyzed (Participants) | 29 | 30 | 30
participants tested positive for ADA
  Screening | 0 | 0 | 1
  End of study | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were evaluated and recorded during the 63 days of the clinical study.
Arm/Group | Zutrab® (Bevacizumab Richmond) | Avastin® | Cizumab®
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 12/29 | 13/30 | 10/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zutrab® (Bevacizumab Richmond) (N=29) | Avastin® (N=30) | Cizumab® (N=30)
Abdominal pain (Gastrointestinal disorders) | 6 (6) | 5 (6) | 4 (4)
Blurry vision (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 4 (5) | 1 (1) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 7 (7) | 6 (6) | 3 (3)
Vomiting (Gastrointestinal disorders) | 4 (4) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-08): https://cdn.clinicaltrials.gov/large-docs/48/NCT03919448/Prot_SAP_000.pdf